CLINICAL TRIAL: NCT05021094
Title: A Multi-center Clinical Study on the Efficacy and Safety of Kuntai Capsule Alone and in Combination With Hormones in the Treatment of Early-onset Hypoovarian Function
Brief Title: Clinical Observation on Kuntai Capsule in Treating Early-onset Ovarian Hypofunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yuquan Zhang, Director of Obstetrics and Gynaecology, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHNantong-POI
Record Dates: First submitted 2021-08-04; First posted 2021-08-25 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Primary Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — kuntai capsule; femoston; Estradiol; Dydrogesterone

STUDY DESIGN:
Intervention Model Description: Subclinical POI and POI patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: blind experiment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- POI patients who taking Kuntai capsule (Experimental): Patients in this group will take Kuntai capsule orally, 4 capsules each time, 3 times a day, and take the medicine for 3 courses.
  Interventions: Drug: Kuntai Capsule
- POI patients who accepting hormone therapy (Active Comparator): The estrogen and progesterone sequential regimen was adopted. The drug was estradiol tablets/estradiol didroxyprogesterone tablets (Femoston). Red tablets (estradiol, 2mg/d) were taken in the first 14 days, and gray tablets (estradiol, 2mg/d, dydrogesterone,10 mg/d) were taken in the last 14 days. 28 days was a course of treatment, and 3 courses of treatment were taken.
  Interventions: Drug: Femoston
- POI patients who taking Kuntai capsule combined with hormone therapy (Experimental): Kuntai capsule was taken at the same dose as Kuntai group on the basis of hormone therapy for 3 courses.
  Interventions: Drug: Kuntai Capsule; Drug: Femoston
- Subclinical POI patients who taking Kuntai capsule (Experimental): Subclinical POI patients in this group which with Kuntai capsule intervention. This group is a self-controlled experiment before and after treatment
  Interventions: Drug: Kuntai Capsule

INTERVENTIONS:
Drug: Kuntai Capsule — The instructions is pointed that each Kuntai capsule is 0.5g and the usage of Kuntai capsule is oral taking 4 capsules each time, 3 times a day, and 4 weeks is a course of treatment. The patients will taking 3 courses of treatment in this study.
  Other Names: Kuntai Jiaonang
  Arms: POI patients who taking Kuntai capsule; POI patients who taking Kuntai capsule combined with hormone therapy; Subclinical POI patients who taking Kuntai capsule
Drug: Femoston — The estrogen and progesterone sequential regimen was adopted. The Femoston was contain estradiol tablets and estradiol didroxyprogesterone tablets. Red tablets (estradiol, 2 mg/d) were taken in the first 14 days, and gray tablets (estradiol, 2 mg/d, dydrogesterone,10 mg/d) were taken in the last 14 days. 28 days was a course of treatment, and three courses of treatment were taken. The patients will taking 3 courses of treatment in this study.
  Other Names: Complex Packing Estradiol Tablets/Estradiol and Dydrogesterone Tablets
  Arms: POI patients who accepting hormone therapy; POI patients who taking Kuntai capsule combined with hormone therapy

SUMMARY:
To evaluate the efficacy and safety of Kuntai capsule alone or combined with hormone therapy in improving ovarian function in POI patients (including subclinical stage).

DETAILED DESCRIPTION:
The study is expected to be conducted between 2021.08 and 2023.12.120 subjects with early-onset ovarian insufficiency will be randomly assigned to trial, control, or combination groups using a computer-generated randomization table.By comparing the data of primary efficacy indexes, secondary efficacy indexes and safety indexes before and after medication, The principal investigator will write and publish the paper.

ELIGIBILITY:
Inclusion Criteria:

1. The women aged <40 years old.
2. Serum basal follicle stimulating hormone (FSH) level ≥15 IU/L at least twice inspection (two occasions >4 weeks apart). Rare menstruation or menopause for at least 4 months.
3. Individuals meeting the above criteria who voluntarily consented to study participation.

Exclusion Criteria:

1. Pregnant and lactating patients;
2. Patients with endometriosis, adenomyosis, endometrial lesions (submucous fibroids, endometrial polyps, etc.), hysteromyoma > 4cm or hysterectomy;
3. Patients with known or suspected breast cancer history and estrogen-dependent malignant tumor;
4. Patients with personal history of venous thromboembolism (VTE) or high risk of VTE (including body mass index > 30 kg/m2, smoking and family history of thrombosis);
5. Patients with porphyria;
6. Patients with serious primary diseases or mental illness such as cardiovascular, liver, kidney and hematopoietic system;
7. Patients who are participating in other clinical trials or have participated in other clinical trials in the past three months;
8. Patients who suspect or have a history of alcohol and drug abuse;
9. Patients who are known to be allergic to the test drugs or their components;
10. The researchers determined that patients are not suitable for this trial.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Follicle-stimulating hormone (FSH) | Baseline, 3 months, 6 months
  Changes of the level of FSH before and after treatment
Kupperman Score | Baseline, 3 months, 6 months
  Changes of the Kupperman score before and after treatment，Kupperman Score ranges from 0 to 69, with the smaller the score, the better off the subject

SECONDARY OUTCOMES:
Luteinizing hormone (LH) | Baseline, 3 months, 6 months
  Changes of the level of LH before and after treatment
Estradiol hormone (E2) | Baseline, 3 months, 6 months
  Changes of the level of Estradiol hormone before and after treatment
Antral follicle count (AFC) | Baseline, 3 months,
  Changes of the AFC before and after treatment
anti-Müllerian hormone (AMH) | Baseline, 3 months,
  Changes of the level of AMH before and after treatment
The peak systolic blood flow velocity （PSV） | Baseline, 3 months,
  The peak systolic blood flow velocity before and after treatment was assessed by vaginal B ultrasound
The end-diastolic blood flow velocity（EDV） | Baseline, 3 months,
  The uterine artery end-diastolic blood flow velocity before and after treatment was assessed by vaginal B ultrasound
Uterine artery resistance index（RI） | Baseline, 3 months,
  The uterine artery resistance index before and after treatment was assessed by vaginal B ultrasound
Proportion of patients with normal menstruation | Baseline，3 months, 6 months, 9 months
  To measure the ratio of patients have normal menstruation after treatment
Pregnancy situation | 6 months
  To ask the patient if there is pregnancy (for patient who has pregnancy need)

CONTACTS AND LOCATIONS:
Overall Officials: Yuquan Zhang, Professor, Principal Investigator — Affiliated Hospital of Nantong University
Locations (6):
- China (6):
  - Hai'an People's Hospital, Hai’an, Jiangsu
  - Hai'an Hospital of traditional Chinese Medicine, Huai'an, Jiangsu
  - Nantong First People's Hospital, Nantong, Jiangsu
  - Nantong Hospital of Traditional Chinese Medicine, Nantong, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Rugao Boai Hospital, Ru'gao, Jiangsu

IPD SHARING:
Plan to Share IPD: No
Not planning sharing at present.

DOCUMENTS (2):
  • Study Protocol (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT05021094/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT05021094/SAP_001.pdf